CLINICAL TRIAL: NCT03040778
Title: Pentoxifylline and Tocopherol (PENTO) in the Treatment of Medication-related Osteonecrosis of the Jaw (MRONJ): A Prospective, Randomized Controlled Trial to Evaluate a Novel Non-operative Treatment
Brief Title: Pentoxifylline and Tocopherol (PENTO) in the Treatment of Medication-related Osteonecrosis of the Jaw (MRONJ)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Alabama at Birmingham (Other); New York Center for Orthognathic and Maxillofacial Surgery (Unknown); University of Michigan (Other)
Responsible Party: Principal Investigator, Jasjit Dillon, Professor & Chief, Program Director, Oral & Maxillofacial Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004779
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Medication-related Osteonecrosis of the Jaw; Bisphosphonate-related Osteonecrosis of the Jaw; Avascular Necrosis
Keywords: MRONJ; BRONJ
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw; Osteonecrosis | interventions — Pentoxifylline; Tocopherols; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care + PENTO (Experimental): The current standard of care for MRONJ as outlined by the American Association of Oral and Maxillofacial Surgeons position paper based on stage of disease (Ruggiero 2014) AND PENTO regimen consisting of 400mg pentoxifylline (PTX) and 400IU tocopherol twice-daily PO for a total of 800mg/day PTX and 800 IU/day tocopherol
  Interventions: Drug: Pentoxifylline; Drug: Tocopherol
- Standard of Care (Placebo Comparator): The current standard of care for MRONJ as outlined by the American Association of Oral and Maxillofacial Surgeons position paper based on stage of disease (Ruggiero 2014). Placebo drugs to be taken in the control group 2 pills BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline is a commonly used medication for muscle pain associated with peripheral artery disease. It is a methylated xanthine derivative that improves peripheral blood flow, flexibility of red blood cell membranes, microcirculation, and tissue oxygenation and reduces viscosity of blood.
  Other Names: Pentoxifylline SR; Trental; Oxpentifylline
  Arms: Standard of Care + PENTO
Drug: Placebo — Placebo tablets
  Arms: Standard of Care
Drug: Tocopherol — Tocopherol (vitamin E) impairs tissue fibrosis and is a potent oxygen radical scavenger that may reduce damage caused by free radicals impacting necrosis.
  Other Names: Vitamin E
  Arms: Standard of Care + PENTO

SUMMARY:
The overall purpose of this project is to answer the following clinical question: Among Medication-Related Osteonecrosis of the Jaw (MRONJ) patients, do those who are treated with the Pentoxifylline and Tocopherol (PENTO) regimen and standard of care, when compared to those treated with standard of care alone, have decreased areas of exposed bone after one year of treatment?

DETAILED DESCRIPTION:
HYPOTHESES

HA: Among patients with MRONJ, after 12 months of treatment with PENTO, the area of exposed bone in the PENTO group will be different than the area of exposed bone in the standard therapy group.

H0: Among patients with MRONJ, after 12 months of treatment with PENTO, the area of exposed bone in the PENTO group will equal the area of exposed bone in the standard therapy group.

SPECIFIC AIMS

To determine if the PENTO regimen in addition to the standard of care treatment for MRONJ significantly reduces the area of exposed bone compared to standard of care alone. Standard of care is defined as the clinical guidelines of the 2014 AAOMS Position Paper on Medication-Related Osteonecrosis of the Jaw (MRONJ)

1. Challenges: Identifying patients with Stage 1, 2, 3 MRONJ who will be compliant with therapy and available for follow-up. Measuring greatest anterior-posterior and superior-inferior dimensions to calculate area. Ensuring patient safety with interim analyses and an appropriate stopping protocol.
2. Approach: The investigators will treat patients with Stage 1, 2, 3 MRONJ with either PENTO as an adjunct to the standard of care or standard of care alone with placebo.

Impact: >6 million patients in the US are at risk for MRONJ. If proven to successfully treat MRONJ, the trial would establish a non-operative treatment option for successful management of MRONJ with potential for significant decreased morbidity for the patient.

SAMPLE

The sample will be derived from the population of patients who present to a participating trial site for management of MRONJ during the trial's enrollment period. To be included in the trial a patient must meet the criteria listed below. If a patient is excluded from the trial the reason will be documented for the study's record as well as basic demographic data, MRONJ staging, risk medications, indication for and use of antiresorptive and antiangiogenic medications and area of exposed bone will be collected.

RANDOMIZATION

A stratified permuted-block randomization will be used to allocate patients to treatment. This method ensures balanced allocations to achieve approximately the preset treatment allocation ratio of 1:1 and avoids predictability of future assignments. Strata will be constructed for the prognostic variables of initial MRONJ stage (1,2,3) and antiresorptive therapy (bisphosphonate vs. denosumab/RANK-L inhibitor). Within each strata, block sizes of 2 and 4 will be used to randomize patients to PENTO + standard of care or to standard of care with placebo alone with randomization of treatment sequence to meet the 1:1 allocation ratio within each block.

A computer-generated list of random allocations will be prepared for each strata. The allocation sequence will be concealed from the researcher enrolling and assessing participants in sequentially numbered, opaque, sealed and stapled envelopes. Corresponding envelopes will be opened only after the enrolled participants complete

DATA MANAGEMENT AND ANALYSIS

The primary analysis of interest is the association between treatment group and area of exposed bone. The primary analysis will be a repeated measures analysis of variance (ANOVA) with one within subject (time) factor and one between subject (treatment) factor will be completed for A = area based upon Dap and Dsi and geometric shape of the lesion. If outcomes do not meet assumptions then non-parametric analogues will be used.

SAMPLE SIZE ESTIMATE

alpha = 0.05, beta = 0.10, Anticipated drop-out rate = 30%

A stratified permuted- block randomization will be used to allocate patients to treatment. Intention to treat to include all subjects as randomized to treatment (detailed on page 3 of the application). If a patient drops out or is withdrawn prior to 12-month treatment endpoint, the last observation carried forward (LOCF) will be included in analysis. In addition, patients "as treated" (patient received incorrect treatment) or "as protocol" (doesn't include patient dropouts or withdrawals) will be analyzed to evaluate effectiveness of the treatment. To detect a relative change in primary outcome ≥20% with the above parameters, a minimum sample of 44 patients in each study arm is required (total n=88).

The investigators deemed that an improvement of ≥20% by the intervention group compared to the control group in decreased bone exposure to be clinically significant. There is no consensus in the current literature on a clinically significant difference between the control and treatment arms. However, if the study is powered for the outcomes expected based on current literature, a difference of 50% between arms would only require 7 patients per arm. Therefore the investigators believe the study to be overpowered to ensure the statistical analysis would remain significant if the suspected success of the PENTO regimen is not true.

STOPPING RULES

Because this is an investigational use of pentoxifylline and the benefits of PENTO in MRONJ are not presently established, interim analyses (p=.001) will be performed at 3 and 6 months. If the trial is stopped after an interim analysis for proven benefit, the trial will be converted to an open trial and the patients will be followed for the entire 12-month treatment period, or until they achieve complete mucosal coverage.

Patient withdrawal from study criteria include:

* A serious adverse event related to the trial medication.
* Patient becomes pregnant.
* Any relevant deterioration in the health of the subject (AEs, vital signs, ECG, laboratory parameters).
* Clinically relevant change in vital signs if technical failure

OVERSIGHT RESPONSIBILITIES

Oversight of the trial is provided by the Principal Investigator (PI) Dr. Dillon and Co- Investigators (Co-I) Dr. Ruggiero, Dr. Morlandt, and Dr. Ward.

MONITORING PROCEDURES

Drs. Dillon, Ruggiero, Morlandt, and Ward assure that informed consent is obtained prior to performing any research procedures, that all subjects meet eligibility criteria, and that the study is conducted according to the IRB-approved research plan. Blinded study data are accessible at all times for the PI and Co-investigators to review. All four investigators will review study conduct including accrual, drop-outs, and protocol deviations on a quarterly basis. In addition, the investigators will review adverse events (AEs) individually real-time and in aggregate on a monthly basis. Last, the investigators will review serious adverse events (SAEs), dose limiting toxicities, and any other specific intervention complications in real-time. The PI ensures all protocol deviations, AEs, and SAEs are reported to the FDA, DSMB and IRB according to the applicable regulatory requirements.

COLLECTION AND REPORTING OF SAEs AND AEs

For this study, the following standard AE definitions are used:

Adverse event (AE): Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.

Serious Adverse Event: Any AE that results in any of the following outcomes:

* Death
* Life-threatening
* Event requiring inpatient hospitalization or prolongation of existing hospitalization
* Persistent or significant disability/incapacity

AEs are graded according to the following scale:

* Mild: An experience that is transient & requires no special treatment or intervention.
* Moderate: An experience that is alleviated with simple therapeutic treatments.
* Severe: An experience that requires therapeutic intervention. The experience interrupts usual daily activities.

The study uses the following AE attribution scale:

* Not related: The AE is clearly not related to the study
* Possibly related: An event that follows a reasonable temporal sequence from the initiation of study procedures, but that could readily have been produced by a number of other factors.
* Related: The AE is clearly related to the study procedures.

SAEs and specific procedure-associated AEs are reported to the University of Washington IRB and DSMB within 24 hours. In addition, all AEs are reported according to the University of Washington IRB AE reporting guidelines.

MANAGEMENT OF RISKS TO SUBJECTS

Expected AEs associated with the Pentoxifylline and Tocopherol include: Dizziness, headache, nausea, vomiting, indigestion, flushing, angina, palpitations, hypersensitivity, itchiness, rash, hives, bleeding, hallucinations, arrhythmias, aseptic meningitis

AE Management

If any unanticipated problems related to the research involving risks to subjects or others happen during the course of this study (including SAEs) these will be reported to the IRB in accordance with University of Washington Human Subjects Division (HSD) protocols and the DSMB. AEs that are not serious but that are notable and could involve risks to subjects will be summarized in narrative or other format and submitted to the IRB and DSMB at the time of continuing review.

DATA SAFETY AND MONITORING (DSMB) ANALYSIS PLAN

The Analysis for safety (AEs) will be conducted at a minimum of 3 and 6 months. However, depending upon recruitment the analysis of safety will be as follows when:

10, 20, 30, 40, 60, 80, 100 patients have completed 3 months of follow up.

Patient withdrawal criteria include:

* A serious adverse event related to the trial medication.
* Patient becomes pregnant.
* Any relevant deterioration in the health of the subject (AEs, vital signs, ECG, laboratory parameters).
* Clinically relevant change in vital signs if technical failure can be excluded and result is confirmed by at least 1 additional measurement.

PLAN FOR DATA MANAGEMENT

Compliance of regulatory documents and study data accuracy and completeness will be maintained through an internal study team quality assurance process.

Confidentiality throughout the trial is maintained by the previously described study-specific confidentiality procedures. DATA will be stored as de-identified on a REDCap database which will be password protected and only accessible by study members.

INFORMED CONSENT/ETHICAL CONSIDERATIONS

Quality and integrity of the research will be ensured through data safety monitoring and informed patient consent for participation. Enrollment will be done by the study coordinator at each site not the participating surgeon. Other than the UW study coordinator the other coordinators will be research students participating in the trial. The research will be independent and impartial, and key study personnel directly involved in patient care will be blinded to the treatment. Informed consents to be obtained from patients will state the overall purpose of the study, alternatives to participation, and any direct and indirect risks/benefits from participation. All patient literature and consents will be written at an 8th grade reading level. The confidentiality and anonymity of the research respondents and patient health information will be respected. IRB approvals will be obtained at all study sites prior to beginning any research activities. The individual study site IRBs will determine if it is appropriate to pursue an expanded access Investigational

ELIGIBILITY:
Inclusion Criteria:

1. Stage 1, 2, or 3 MRONJ as defined by the AAOMS Position Paper on Medication-Related Osteonecrosis of the Jaw-2014 Update (Ruggiero 2014).
2. History of exposure to antiresorptive medications such as bisphosphonates or RANK-L inhibitors
3. Absence of tumor in the jaw at the time of recruitment
4. Patients with the capacity to give informed consent

Exclusion Criteria:

1. Patients with history of external radiation therapy to the jaws
2. Patients who underwent any surgical intervention for MRONJ in the past 4 months
3. Patients with past microvascular reconstruction of the head and neck
4. Patients with an expected survival less than 1 year
5. Patients with allergy or hypersensitivity to pentoxifylline, xanthines, or tocopherol
6. Patients with planned invasive dental procedure in the next year
7. Patients taking oral anticoagulants
8. Patients with known hemorrhagic and coagulation disorder
9. Patients with a vitamin K deficiency due to any cause
10. Female patients who are pregnant or lactating
11. Patients with history of serious bleeding or extensive retinal hemorrhage
12. Patients with ischemic heart diseases, including, but not limiting, recent myocardial infarction
13. Patients with serious cardiac arrhythmia
14. Patients with severe liver disease
15. Patients with severe renal failure (Creatinine clearance <30 mL/min)
16. Patients with diagnosed hypotension
17. Patients taking CYP1A2 inhibitors (e.g. ciprofloxacin, fluvoxamine)
18. Diagnosis of MRONJ with no exposed bone
19. Patient cannot tolerate impressions of exposed bone in a clinical setting, if needed.
20. There is a change in the patient's clinical presentation (tooth extraction, sequestrectomy) from alginate impression, if impression is indicated.
21. Any other situation or condition that, in the opinion of the INVESTIGATOR, may interfere with optimal PARTICIPATION in the study
22. • Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
23. Patients who are taking additional vitamin E, or you will confirm they will stop taking vitamin E if they decide to enroll in this study.
24. Patients who are taking oral anticoagulant medications.
25. Discuss with patients taking aspirin and other supplements/medications that impact coagulation to determine if the study is a good fit, and will exclude an individual whose situation or condition may interfere with safe participation in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Bone exposure area (mm^2) | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  The primary lesion's area of exposed bone will be estimated by measuring the greatest anterior-posterior and superior-inferior dimensions in millimeters (mm) of the site with the largest area of exposed bone present at the time of study enrollment.
  If there are multiple areas of exposed bone in a single patient, the site with the largest sum of linear anterior-posterior and superior-inferior dimensions will be included in the study.

SECONDARY OUTCOMES:
Change in MRONJ Stage | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  MRONJ staging based on AAOMS Position paper staging criteria (Stage 0,1,2,3)
Change in Pain | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  Visual analogue scale (VAS) measure of pain. A 100 mm scale will be used with 0 = no pain and 100 = worst pain ever. The patient will be asked to indicate their level of on the VAS.
Change in osseous anterior-posterior linear dimension on orthopantomogram | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  Radiographic analysis. Greatest anterior-posterior linear dimension of osseous changes. A 5mm ball bearing will be used to standardize the measurement.
Change in osseous superior-inferior linear dimension on orthopantomogram | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  Radiographic analysis. Dsi= Greatest superior-inferior linear dimension of osseous changes. A 5mm ball bearing will be used to standardize the measurement.
Change in osseous area on orthopantomogram | 0 months, 1 month, 3 months, 6 months, 9 months, 12 months
  Radiographic analysis. Change in area of osseous change. Will be according to the above formulae for shape; rectangle, circle, ellipse for the orthopantomogram imaging. A 5mm ball bearing will be used to standardize the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Jasjit Dillon, DDS, MBBS, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - New York Center for Orthognathic and Maxillofacial Surgery, Lake Success, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delanian S, Chatel C, Porcher R, Depondt J, Lefaix JL. Complete restoration of refractory mandibular osteoradionecrosis by prolonged treatment with a pentoxifylline-tocopherol-clodronate combination (PENTOCLO): a phase II trial. Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):832-9. doi: 10.1016/j.ijrobp.2010.03.029. Epub 2010 Jul 16. PMID 20638190
- [Background] Delanian S, Depondt J, Lefaix JL. Major healing of refractory mandible osteoradionecrosis after treatment combining pentoxifylline and tocopherol: a phase II trial. Head Neck. 2005 Feb;27(2):114-23. doi: 10.1002/hed.20121. PMID 15641107
- [Background] Epstein MS, Wicknick FW, Epstein JB, Berenson JR, Gorsky M. Management of bisphosphonate-associated osteonecrosis: pentoxifylline and tocopherol in addition to antimicrobial therapy. An initial case series. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Nov;110(5):593-6. doi: 10.1016/j.tripleo.2010.05.067. PMID 20955948
- [Background] Magremanne M, Reychler H. Pentoxifylline and tocopherol in the treatment of yearly zoledronic acid-related osteonecrosis of the jaw in a corticosteroid-induced osteoporosis. J Oral Maxillofac Surg. 2014 Feb;72(2):334-7. doi: 10.1016/j.joms.2013.06.188. Epub 2013 Jul 25. PMID 23891014
- [Background] McLeod NM, Pratt CA, Mellor TK, Brennan PA. Pentoxifylline and tocopherol in the management of patients with osteoradionecrosis, the Portsmouth experience. Br J Oral Maxillofac Surg. 2012 Jan;50(1):41-4. doi: 10.1016/j.bjoms.2010.11.017. Epub 2011 Jan 19. PMID 21247671
- [Background] Ruggiero SL, Dodson TB, Fantasia J, Goodday R, Aghaloo T, Mehrotra B, O'Ryan F; American Association of Oral and Maxillofacial Surgeons. American Association of Oral and Maxillofacial Surgeons position paper on medication-related osteonecrosis of the jaw--2014 update. J Oral Maxillofac Surg. 2014 Oct;72(10):1938-56. doi: 10.1016/j.joms.2014.04.031. Epub 2014 May 5. PMID 25234529
- [Background] Delanian S, Lefaix JL, Maisonobe T, Salachas F, Pradat PF. Significant clinical improvement in radiation-induced lumbosacral polyradiculopathy by a treatment combining pentoxifylline, tocopherol, and clodronate (Pentoclo). J Neurol Sci. 2008 Dec 15;275(1-2):164-6. doi: 10.1016/j.jns.2008.08.004. Epub 2008 Sep 19. PMID 18804790
- [Background] Delanian S, Porcher R, Rudant J, Lefaix JL. Kinetics of response to long-term treatment combining pentoxifylline and tocopherol in patients with superficial radiation-induced fibrosis. J Clin Oncol. 2005 Dec 1;23(34):8570-9. doi: 10.1200/JCO.2005.02.4729. Epub 2005 Oct 31. PMID 16260695
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376